CLINICAL TRIAL: NCT00582556
Title: Phase II Trial of Zometa on Bone Mineral Density on Patients With Stage D Prostate Cancer Undergoing Androgen Ablation Therapy
Brief Title: Zometa on Bone Mineral Density in Prostate Cancer Patients Undergoing Androgen Ablation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO02807; CO02807 (Other: University of Wisconsin Carbone Cancer Center); 2003-057 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE (Other: UW Madison); NCI-2011-00712 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2014-06

CONDITIONS: Prostate Cancer
Keywords: bone mineral density
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): GnRH analogue 3-mo depot - q3 months for 1 yr and Zometa 4 mg IV over 15 min x 1, given 7 days prior to beginning androgen deprivation therapy
  Interventions: Drug: Zometa
- 2 (Active Comparator): GnRH analogue 3-mo depot - q3 months for 1 yr and Zometa 4 mg IV over 15 min x 1, given at mo 6
  Interventions: Drug: zometa
- 3 (Active Comparator): GnRH analogue 3-mo depot - q3 months for 1 yr and Zometa 4 mg IV over 15 min, given monthly x 6 months, beginning in month 6.
  Interventions: Drug: Zometa

INTERVENTIONS:
Drug: Zometa — GnRH analogue 3-mo depot - q3 months for 1 yr and Zometa 4 mg IV over 15 min x 1, given 7 days prior to beginning androgen deprivation therapy
  Other Names: zoledronic acid; lupron; zolodex
  Arms: 1
Drug: zometa — GnRH analogue 3-mo depot - q3 months for 1 yr andZometa 4 mg IV over 15 min x 1, given at mo 6
  Other Names: zoledronic acid; lupron; zolodex
  Arms: 2
Drug: Zometa — GnRH analogue 3-mo depot - q3 months for 1 yr and Zometa 4 mg IV over 15 min, given monthly x 6 months, beginning in month 6.
  Other Names: zolodronic acid; lupron; zolodex
  Arms: 3

SUMMARY:
The purpose of this research is to determine the effect of timing of Zometa® administration on bone mineral density of the lumbar spine and femoral neck in men undergoing androgen deprivation therapy for prostate adenocarcinoma. In addition, the researchers will also determine the effects of treatment with Zometa® on peripheral blood markers of bone turnover, on peripheral blood gd T-cell frequencies and function, and to determine if the above treatments elicit prostate antigen-specific IgG immune responses. The effects of the above treatments on serial serum PSA measurements will also be examined.

DETAILED DESCRIPTION:
Castration by GnRH agonist therapy with or without androgen antagonists has been a mainstay for advanced prostate cancer. One of the most significant side effects of the use of androgen ablative therapies has been a decrease in bone mineral density, potentially placing patients at greater risk of osteoporosis and bone fractures. It is prudent to anticipate this adverse effect of therapy and to minimize its severity with appropriate and timely pharmacologic intervention. Zometa is a bisphosphonates and bisphosphonates are effective inhibitors of osteoclastic bone resorption. Recent studies have shown that other bisphosphonates were able to reduce the bone loss observed after 24 and 48 weeks of treatment with a GnRH analogue. An unanswered question remains, however, in how frequently these agents should be employed in clinical practice.

This is a three-arm randomized trial of Zometa® on bone mineral density in subjects with stage D prostate cancer undergoing androgen ablation therapy. If subjects are enrolled in Arm 1, the GnRH analogue would be administered every 3 months for 1 year. Four milligrams of Zometa® would be administered IV over 15 minutes 7 days prior to beginning androgen deprivation therapy. If subjects are enrolled in Arm 2, the GnRH analogue would be administered every 3 months for one year, and 4 mg of Zometa® would be administered IV over 15 minutes at month 6. If subjects are enrolled in Arm 3, the GnRH analogue is administered every 3 months for 1 year, with 4 mg of Zometa® administered IV over 15 minutes monthly for 6 months, beginning at month 6.

ELIGIBILITY:
Inclusion Criteria:

* Must have a histologic diagnosis of adenocarcinoma of the prostate.
* For patients without clinical metastasis treated by surgery, serum PSA values must be > 0.2 ng/ml by two measurements at least two weeks apart. In patients treated with ablative radiation therapy without clinical metastasis, three consecutive increases in serum PSA must be documented, with at least a one-month interval between values with the final PSA > 2ng/m as evidence of biochemical PSA failure. P
* Patients who have not had prior primary therapy such as radiation or surgery, are required to have a detectable PSA of at least 0.2 ng/ml.
* Patients with evidence of metastatic disease are eligible irrespective of serum PSA level.
* Prior history of a second malignancy is allowed if treated with curative intent and patient has been free of disease greater than five years
* ECOG performance status of < 2.

Exclusion Criteria:

* Prior treatment with a GnRH analogue or anti-androgen.
* Evidence of immunosuppression or have been treated with immunosuppressive therapy, such as chemotherapy, chronic treatment dose corticosteroids, or radiation therapy to bones, within 6 months of study enrollment
* Current or treatment within 4 weeks with estrogen or estrogenic agents (including herbal compound PC-SPES)
* Current or treatment within 4 weeks with herbal compounds for prostate cancer such as PC-SPES or saw palmetto
* Current or treatment within 4 weeks with megestrol
* Current or prior treatment with a bisphosphonate, calcitonin, or other bone resorptive/anabolic agents
* Current use of oral corticosteroids or any such use within the past 6 months
* Current use of potentially bone-toxic anticonvulsants (phenytoin, or carbamazepine)
* History of orchiectomy
* Hypocalcemia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-04; Primary Completion 2011-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McNeel, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at the University of Wisconsin Carbone Cancer Center from April 2003 until March 2011.
Pre-assignment Details: Of the 44 subjects enrolled, one withdrew from the study prior to receiving any study treatment. As a result there were 43 subjects who received at least one dose of study medication.
Groups:
- Zometa Given 7 Days Prior to Beginning ADT: GnRH analogue 3-mo depot - q3 months for 1 yr and Zometa 4 mg IV over 15 min x 1, given 7 days prior to beginning androgen deprivation therapy
- Zometa Given at Month 6: GnRH analogue 3-mo depot - q3 months for 1 yr and Zometa 4 mg IV over 15 min x 1, given at mo 6
- Zometa Given Monthly x 6 Months: GnRH analogue 3-mo depot - q3 months for 1 yr and Zometa 4 mg IV over 15 min, given monthly x 6 months, beginning in month 6.
Period: Overall Study
Arm/Group | Zometa Given 7 Days Prior to Beginning ADT | Zometa Given at Month 6 | Zometa Given Monthly x 6 Months
Started | 14 | 15 | 14
Completed | 14 | 14 | 12
Not Completed | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zometa Given 7 Days Prior to Beginning ADT | Zometa Given at Month 6 | Zometa Given Monthly x 6 Months | Total
Number analyzed (Participants) | 14 | 15 | 14 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 10 | 32
  >=65 years | 3 | 4 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 14 | 15 | 14 | 43
Gleason Score of 8 or more [Number; unit: participants] — The Gleason score is a sum of two scores--each ranging between 1 and 5--provided by the pathologist who examines the cancer under the microscope. When you add the 2 scores you get the Gleason sum which ranges from 2-10: 2 looking basically like a normal prostate and 10 looking extremely aggressive.
  participants | 3 | 4 | 8 | 15
Participants with evidence of osteopenia/osteoporosis [Number; unit: participants] | 6 | 4 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Who Had Either an Increase or Decrease on Bone Mineral Density of the Lumbar Spine and Femoral Neck in Men Undergoing Androgen Deprivation Therapy for Prostate Adenocarcinoma.
Description: Effects on bone mineral density were measured at four locations at six month intervals for 24 months.
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- Zometa Given Monthly, Months 6-11: GnRH analogue 3-mo depot - q3 months for 1 yr and Zometa 4 mg IV over 15 min, given monthly x 6 months, beginning in month 6.
Arm/Group | Zometa Given 7 Days Prior to Beginning ADT | Zometa Given at Month 6 | Zometa Given Monthly, Months 6-11
Number analyzed (Participants) | 14 | 15 | 15
participants | 14 | 15 | 15

2. Secondary Outcome: The Number of Subjects Who Had a Significant Increase of Peripheral Blood Markers of Bone Turnover.
Description: Serum bone-specific alkaline phosphatase was collected as the blood marker of bone turnover.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Zometa Given 7 Days Prior to Beginning ADT | Zometa Given at Month 6 | Zometa Given Monthly, Months 6-11
Number analyzed (Participants) | 14 | 15 | 15
participants | 0 | 0 | 0

3. Secondary Outcome: Number of Subjects Had a Significant Change in Immune Markers.
Description: Immune markers were measured by isolating gamma-delta T cells one month after treatment with zoledronic acid.
Time Frame: 2 Years
Measure: Number; unit: participants
Arm/Group | Zometa Given 7 Days Prior to Beginning ADT | Zometa Given at Month 6 | Zometa Given Monthly, Months 6-11
Number analyzed (Participants) | 14 | 15 | 15
participants | 0 | 0 | 0

4. Secondary Outcome: Number of Subjects With Decreases in Prostate Specific Antigen (PSA) After Zoledronic Acid Prior to Beginning Androgen Deprivation Therapy
Description: PSA response was measured by observing the serum PSA one week after beginning zoledronic acid and prior to beginning androgen deprivation therapy.
  Arm 2 and Arm 3 were not able to be assessed for this endpoint as all subjects were on androgen deprivation prior to receiving zoledronic acid.
Time Frame: 2 Years
Measure: Number; unit: participants
Groups:
- Zometa Given 7 Days Prior to Beginning ADT: Gonadotropin releasing hormone (GnRH) analogue 3-mo depot - q3 months for 1 yr and Zometa 4 mg IV over 15 min x 1, given 7 days prior to beginning androgen deprivation therapy
Arm/Group | Zometa Given 7 Days Prior to Beginning ADT | Zometa Given at Month 6 | Zometa Given Monthly, Months 6-11
Number analyzed (Participants) | 14 | 0 | 0
participants | 0 |  |

ADVERSE EVENTS:
Time Frame: 6 years and 7 months
Arm/Group | Zometa Given 7 Days Prior to Beginning ADT | Zometa Given at Month 6 | Zometa Given Monthly x 6 Months
Serious Adverse Events (participants affected / at risk) | 2/14 | 2/15 | 2/15
Other Adverse Events (participants affected / at risk) | 14/14 | 15/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Zometa Given 7 Days Prior to Beginning ADT (N=14) | Zometa Given at Month 6 (N=15) | Zometa Given Monthly x 6 Months (N=15)
Low Platelets (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0/14 (0)
Creatine phosphokinase (Metabolism and nutrition disorders) | 1 (1) | 0 | 0/14
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0/14
Musculoskeletal/Soft Tissue - Other (Complication of prior hip replacement) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0/14
Chest Pain (non-cardiac and non-pleuritic) (General disorders) | 1 (1) | 0 | 0/14 (0)
Musculoskeletal-Other (fracture) (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0/14
Creatinine (Renal and urinary disorders) | 1 (1) | 0 | 0/14
Infection without neutropenia (Infections and infestations) | 0 | 1 (1) | 0/14
Musculoskeletal-other (shoulder) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0/14
Syncope (fainting) (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Right Hip Replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - abdomen (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Epidural hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary-Other (pneumonia) (Infections and infestations) | 0 | 0 | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zometa Given 7 Days Prior to Beginning ADT (N=14) | Zometa Given at Month 6 (N=15) | Zometa Given Monthly x 6 Months (N=15)
Hot flashes (Endocrine disorders) | 11 (14) | 11 (13) | 11 (14)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (11) | 5 (6) | 3 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (4) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (13) | 3 (3) | 3 (6)
Pain - other (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 4 (8)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain or cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (non-cardiac and non-pleuritic) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (4) | 1 (1) | 6 (8)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (4)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Anorexia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Salivary Gland Changes (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis/pharyngitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Taste Disturbance (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy-sensory (Nervous system disorders) | 4 (4) | 2 (2) | 2 (4)
Mood alteration-depression (Nervous system disorders) | 1 (3) | 0 (0) | 3 (3)
Insomnia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Neurology--other (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (2) | 1 (3) | 1 (1)
Dizziness/Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory Loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mood alteration-anxiety, agitation (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2) | 3 (4) | 1 (1)
Creatinine (Renal and urinary disorders) | 2 (3) | 1 (1) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal/Genitourinary-Other (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 3 (3) | 5 (5) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 2 (2)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (6) | 8 (9) | 7 (12)
Pelvic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
weight gain (Investigations) | 1 (1) | 1 (1) | 2 (3)
Fever (in the absence of neutropenia) (General disorders) | 2 (2) | 0 (0) | 0 (0)
Rigors (chills) (General disorders) | 0 (0) | 1 (2) | 1 (1)
Sweating (diaphoresis) (General disorders) | 1 (1) | 0 (0) | 1 (1)
Constitutional Symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Auditory/Hearing-Other (hearing loss from broken vessel in ear) (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
Infection without neutropenia (Infections and infestations) | 1 (2) | 3 (3) | 3 (4)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Vision - flashing lights/floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Creatine phosphokinase (Investigations) | 1 (3) | 0 (0) | 0 (0)
Hypercalcemia (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Investigations) | 0 (0) | 0 (0) | 1 (1)
Erectile impotence (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Libido (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Low Hemoglobin (Investigations) | 1 (2) | 0 (0) | 0 (0)
Low Leukocytes (Investigations) | 1 (3) | 0 (0) | 0 (0)
Low Platelets (Investigations) | 1 (3) | 0 (0) | 0 (0)
SGOT (AST) (Investigations) | 1 (4) | 0 (0) | 0 (0)
SGPT (ALT) (Investigations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes